CLINICAL TRIAL: NCT06731608
Title: Effectiveness of an Multi-Modal Intervention for Transitions of Care After Lower Limb Fracture
Brief Title: OsteoPorotic fracTure preventION System (OPTIONS) Research Study
Acronym: OPTIONS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: University of Maryland, Baltimore (Other); Hebrew SeniorLife (Other); Patient-Centered Outcomes Research Institute (Other); University of Arkansas (Other); Emory University (Other)
Responsible Party: Principal Investigator, Kumiko O. Schnock, Instructor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024P002736; OFP-2021C3-24922 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2024-12-04; First posted 2024-12-12 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Osteoporosis; Lower Limb Fracture
Keywords: Osteoporosis; Lower Limb Fracture; Post-fracture Care; Fracture Prevention
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Intervention Model Description: A matched-pair cluster randomized controlled trial (RCT) design
Who Masked: Outcomes Assessor
Masking Description: The OsteoPorotic fracTure preventION System (OPTIONS) intervention is a facility-level initiative for Skilled Nursing Facilities (SNFs) and 21 SNF sites will receive the OPTIONS intervention, while 21 SNF sites will serve as a comparator group, receiving enhanced usual care with the Stopping Elderly Accidents, Deaths, and Injuries (STEADI) Toolkit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- OPTIONS intervention (Experimental): OPTIONS is a multimodal intervention approach that includes providing clinical decision support (CDS) for healthcare providers, patients, and their caregivers focused on exercise, nutrition, and bone-enhancing medications using CDS in SNFs that use the same electronic health record system (PointClickCare).
  Interventions: Behavioral: OPTIONS
- Enhanced Usual Care (Active Comparator): Enhanced usual care includes access to the STEADI (Stopping Elderly Accidents, Deaths, and Injuries) toolkit, a fall prevention program from the CDC.
  Interventions: Behavioral: Enhanced usual care

INTERVENTIONS:
Behavioral: OPTIONS — OPTIONS is a multimodal intervention approach that includes providing clinical decision support (CDS) for healthcare providers, patients, and their caregivers focused on exercise, nutrition, and bone-enhancing medications using CDS in SNFs that use the same electronic health record system (PointClickCare).
  Arms: OPTIONS intervention
Behavioral: Enhanced usual care — Enhanced usual care includes access to the STEADI (Stopping Elderly Accidents, Deaths, and Injuries) toolkit, a fall prevention program from the CDC.
  Arms: Enhanced Usual Care

SUMMARY:
Osteoporosis is a disease that weakens bones so the bones may break easily. The risk for osteoporosis increases with age in both women and men. Osteoporosis affects 10 million older adults in the US. Osteoporosis is a common cause of broken bones in the hips and legs. Broken bones can lead to disability, nursing home placement, and death. Because of the dire consequences, a broken hip or leg is one of the most dreaded injuries for older adults. Many studies confirm that a simple regimen of exercise, healthy diet and bone-strengthening medications can improve overall recovery after a broken hip or leg. This regimen can prevent a person from becoming disabled, having future fractures, and even prevent death.

Many older adults have surgery in a hospital after breaking a hip or leg. Then older adults go to a skilled nursing facility (SNF) for rehabilitation. Care in SNFs varies greatly. Some patients do not receive the regimen that the investigators know is most beneficial to improve bone health and recovery. Even patients who get exercise, healthy diet, and bone-strengthening medication in the SNF, may not continue with the regimen once patients go home. Therefore, the investigators want to implement and test OsteoPorotic fracTure preventION System (OPTIONS). OPTIONS is a program that will integrate the regimen into the care that is provided in SNFs and after discharge to the community. OPTONS will provide information about exercise, diet, and bone-strengthening medication. OPTIONS will provide doctors, clinical staff, patients, and care partners with the information these stakeholders need to carry out the best-practice regimen.

The investigators are partnering with PointClickCare, a large cloud-based healthcare software provider, with SNFs and community care sites across the US. The investigators will include 32 SNFs from different US areas. The investigators will flip a coin to assign SNFs to the intervention (OPTIONS) or the control arm (enhanced usual care) of the study. Enhanced usual care is the care that is typically provided in SNFs after a fracture and adding information about a publicly available fall prevention toolkit. The investigators are using an "implementation science" approach that requires the investigators to get input from the OPTIONS study's vast stakeholder community throughout the study. The OPTIONS study's stakeholders include patients, care partners, clinicians, and professional organizations.

The research question is, can using OPTIONS in SNFs and in the community after discharge improve physical function and quality of life in older people in the year after a hip or leg fracture? The investigators are measuring patient-reported outcomes. The investigators will include 1553 patients across the 32 facilities. The investigators have selected outcomes that are important to patients. Specifically, the investigators are measuring patient-reported function and quality of life. The investigators are also measuring patient-reported falls and fractures. The investigators will track the number of patients who die during the study. This study's hypothesis is that patients who receive OPTIONS will report better physical function (i.e., can walk and take better care of themselves) than those who receive enhanced usual care. The investigators also hypothesize that patients that receive OPTIONS will report a better quality of life than those who receive enhanced usual care.

This study will provide sound data about the effectiveness of OPTIONS. OPTIONS could then be spread to other SNFs and community-based programs. This would ensure that all older people receive the right care after a hip or leg fracture.

DETAILED DESCRIPTION:
There are 10 million older adults (65+) with osteoporosis in the United States of America contributing to over 2 million fragility fractures annually that result in disability, nursing home placement, and mortality. Older adults with lower limb fractures receive acute care and surgery in hospital and are discharged within 3-5 days to a skilled nursing facility (SNF) for rehabilitation where care is highly heterogenous. Length of stay in SNF can be 3-12 weeks and offers the ideal setting for initiating evidence-based interventions across the clinical care team and allowing for targeted education for the patient and family. The investigators propose to introduce OsteoPorotic fracTure preventION System (OPTIONS), an integrated multi-modal intervention, with clinical decision support (CDS), for providers, patients, and care partners, to improve uptake of tailored exercise, healthy nutrition, and bone-enhancing medications. The investigators focus on those who were community-dwelling at the time of fracture entering SNFs for rehabilitation and their transitions back to the community. CDS is needed to quickly and easily guide clinicians to the most effective strategies for an individual patient and engage patients and their caregivers in decision-making to ensure that the evidence-based interventions are routinely implemented and sustained in clinical practice within the SNF and across transitions in the community.

The investigators will partner with PointClickCare, a large cloud-based healthcare software provider and with SNFs across the United States to conduct a matched pair cluster randomized controlled trial (SNF as unit of randomization) across 32 SNFs. The purpose of this project is to determine the effectiveness of OPTIONS to improve function and quality of life by increasing uptake and adherence of 3 evidence-based clinical interventions: functional exercises, nutrition, and bone-enhancing medications. The investigators will compare outcomes from 776 older patients with access to OPTIONS in 16 SNFs versus enhanced usual care (n=776 patients in 16 SNFs) in the year after lower limb fracture across transitions of care from SNF to community-based care. The OPTIONS intervention and implementation will be informed by the OPTIONS study's stakeholder community which consists of patients, caregivers, professional and para-professional providers, and professional organizations.

It is critical to use both effectiveness and implementation science aims to maximize rigor in testing OPTIONS' effectiveness and in developing and testing the implementation protocol to produce a widely reproducible product. To ensure successful implementation in a large number of complex care environments (SNF/Community), the investigators will first use the RE-AIM (reach, effectiveness, adoption, implementation, and maintenance) implementation science framework to develop an OPTIONS implementation toolkit during a pilot implementation phase using semi-structured interviews with key stakeholders (SNF staff, patients, and care partners). Based on this qualitative feedback, the investigators will refine the implementation protocol and toolkit for conducting the cluster randomized trial. The investigators will also use RE-AIM to refine the OPTIONS implementation toolkit at the end of the trial with additional qualitative interviews to facilitate widespread dissemination of the OPTIONS intervention.

The study's specific aims are:

Outcome Aim: Evaluate the effectiveness of OPTIONS versus enhanced usual care for improving function and quality of life (primary outcomes) by increasing uptake and adherence of 3 evidence-based clinical interventions: functional exercise, nutrition, and bone-enhancing medications, across SNF and community care transitions in the first year after lower limb fracture. Secondary and tertiary outcomes include self-reported falls and fractures, mortality (secondary outcomes); measures of adherence to the trimodal interventions in the year after lower limb fracture, and primary care follow-up rates after discharge from SNF (tertiary outcomes).

Implementation Aim: Evaluate the effectiveness of the OPTIONS implementation process and adherence during SNF and community care transitions, during the pilot phase and at trial completion, using content analysis of qualitative data from key stakeholders. The investigators will produce an implementation toolkit to facilitate spread beyond project sites that will include tools to address the following: 1) Process evaluation including implementation progress and identification of processes that worked well or need adjustment. 2) Readiness for Implementation checklist. 3) Classification of adoption success using a rating system that will allow future sites to redress ongoing issues after the initial implementation period.

This study will provide reliable evidence about the effectiveness of OPTIONS that could be widely disseminated to other SNFs providing rehabilitative care and community-based programs to ensure that tailored prevention recommendations and prescriptions are evidence-based and consistent with patients' needs and preferences.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years old
* Community-dwelling at the time of fracture
* Admission to a participating SNF for rehabilitation following a lower limb fragility fracture, including pelvic fractures
* Expected discharge to the community (home or assisted living)

Exclusion Criteria:

* Not English or Spanish speaker
* Admission Brief Interview for Mental Status (BIMS) score 0-7
* SNF length of stay < 7 days
* Regular access to a working telephone or other communication device
* Receiving hospice or end-of-life care

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1344 (Estimated)
Dates: Start 2026-01-16 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Patient-reported function | Discharge from a SNF within four weeks and at six months and twelve months post-SNF discharge (three-time points)
  Daily Activity Scale of the Activity Measure for Post-Acute Care (AM-PAC) Daily Activity Outpatient Short Form (Low Function): The AM-PAC measures a patient's functional ability to perform daily activities, with higher scores indicating greater independence (raw scores range from 6 to 24).
Patient-reported quality of life | Discharge from a SNF within four weeks and at six months and twelve months post-SNF discharge (three-time points)
  Euroqol-5-Dimension Questionnaire-3-Level (EQ-5D-3L): The EQ-5D-3L measures health-related quality of life (Mobility, Self-care, Usual activities, Pain or discomfort, and Anxiety or depression). The best possible health state is represented by score of 1, and the worst possible health state is less than 0.

SECONDARY OUTCOMES:
Number of patients with Falls | Discharge from a SNF within four weeks and at six months and twelve months post-SNF discharge (three-time points)
  Patient self-reported falls: number of falls in the past 6 months
Patient Reported Falls Efficacy | Discharge from a SNF within four weeks and at six months and twelve months post-SNF discharge (three-time points)
  Patient Reported Falls Efficacy: The fall-efficacy scale contains 10 questions on a scale from 1 to 10, with 1 being very confident and 10 being not confident at all. A total score of greater than 70 indicates that the person has a fear of falling.
Number of patients with Fractures | Discharge from a SNF within four weeks and at six months and twelve months post-SNF discharge (three-time points)
  Patient self-reported fractures: number of patients with fractures in the past 6 months
Care Partner Reported Mortality Rate | Six months and twelve months post-SNF discharge (two-time points)
  Care partner reported mortality rate: the number of deaths in the past six months
Function-Mobility | Discharge from a SNF within four weeks and at six months and twelve months post-SNF discharge (three-time points)
  AM-PAC® Basic Mobility Outpatient Short Form (Low Function): The AM-PAC measures a patient's ability to perform basic mobility tasks, with higher scores reflecting greater independence (raw scores range from 6 to 24)
Social Isolation | Discharge from a SNF within four weeks and at six months and twelve months post-SNF discharge (three-time points)
  PROMIS Social Isolation - Short Form 8a: PROMIS Social Isolation - Short Form 8a is an 8-item questionnaire that measures an individual's perception of being socially isolated, feeling excluded, or disconnected from others
Bone Health Behaviors (exercise, nutrition, and bone-enhancing medications) | Discharge from a SNF within four weeks and at six months and twelve months post-SNF discharge (three-time points)
  Self reported questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Denise Orwig, PhD, Principal Investigator — University of Maryland, Baltimore; Patricia Dykes, RN, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - University of Maryland, Baltimore, Department of Epidemiology and Public Health, Division of Gerontology, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No